CLINICAL TRIAL: NCT03150303
Title: Survey About Oral Anticoagulant Peri-procedural Management in Patients Undergoing an Oral Surgery, Implantology or Periodontology
Brief Title: Oral Anticoagulant Peri-procedural Management in Patients Undergoing an Oral Surgery, Implantology or Periodontology
Acronym: PRADICO
Status: Terminated | Type: Observational
Why Stopped: Lack of budget
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bristol-Myers Squibb (Industry); Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: HAO-16007
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2017-04

CONDITIONS: Oral Anticoagulants; Invasive Procedure
Keywords: Periprocedural period; Anticoagulant treatment; Thromboembolic events; Bleeding events
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitamin K Antagonists (VKA): Patients on VKA
- Direct Oral Anticoagulant (DOAC): Patients on OAD

SUMMARY:
Patients receiving long-term oral anticoagulant (defined as duration of treatment of at least 1 month of Direct Oral Anticoagulant (DAOC) or Vitamin K Antagonist (VKA)) and referred for an invasive procedure (oral surgery, implantology or periodontology) to an oral surgeon taking part to the study will be included in this prospective observational study.

The main composite outcome is the occurrence rate of hemorrhagic and/or thromboembolic events during the peri-procedural period (between 5 days before surgery plus 30 days after the invasive procedure).

0. The secondary end-points will consist of identifying risk factors for bleeding during the peri-procedural period, risk factors for thromboembolic events during the peri-procedural period, the peri-procedural management of each treatment (VKA or DOAC), the prescribers involved in the possible change of anticoagulant prescription prior the oral surgery All outcome events will be blindly adjudicated by a central independent adjudication committee.

DETAILED DESCRIPTION:
Manager Centre de Pharmaco-épidémiologie de l'AP-HP

Title Survey about oral anticoagulant peri-procedural management in patients undergoing an oral surgery, implantology or periodontology

Acronym PRADICO

Investigator Coordinator Isabelle MAHE

Number of investigational sites 100

Number of patients 2000

Population Patients receiving oral anticoagulant undergoing an oral surgery, implantology or periodontology

Research calendar Duration of inclusions: 1 year Duration of follow up: 30 days Study duration: 13 months

Selection criteria

Inclusion criteria :

Patients receiving long-term oral anticoagulant (defined as duration of treatment of at least 1 month) and referred for an invasive procedure (oral surgery, implantology or periodontology) to an oral surgeon member of the SFCO (Société Française de Chirurgie Orale) or a periodontologist member of the SFPIO (Société Française de Parodontologie et d'Implantologie Orale) taking part to the study.

Each investigator will include 10 patients treated with long-term DOAC, and 10 consecutive patients treated with long-term VKA. For the DOAC group, inclusion will be continued until the inclusion of 333 patients for each molecule (apixaban, rivaroxaban, edoxaban).

Non-inclusion criteria :

Patients receiving both VKA and antiplatelet agents Patients receiving both direct oral anticoagulant and antiplatelet agents

Objectives

Primary aim:

To assess the composite rate of thromboembolic and bleeding events occurring within the peri-procedural period, in patients on long-term DOAC and VKA and undergoing an oral surgery, implantology or periodontology.

Secondary aims :

* To identify risk factors for bleeding during the peri-procedural period
* To identify risk factors for thromboembolic events during the peri-procedural period
* To describe the peri-procedural management of each treatment (VKA or DOAC)
* To identify prescribers involved in the possible change of anticoagulant prescription prior the oral surgery
* To compare the risk of bleeding on DOAC and on VKA
* To compare the risk of thromboembolic complications on DOAC and on VKA
* To evaluate the net clinical benefit of DOAC compared to VKA treatment

Endpoints

Primary endpoint :

A composite outcome: the occurrence rate of hemorrhagic and/or thromboembolic events during the peri-procedural period.

Secondary endpoints :

* Incidence of bleeding events
* incidence of thromboembolic events
* net clinical benefit of DOAC compared to VKA

Methodology Prospective observational non interventional multicentric cohort study in adult population under long-term anticoagulant treatment (DOAC or VKA) and undergoing an oral, periodontal or implant surgery, by liberal practitioners or oral specialists at hospital.

Statistical analysis The occurrence rate of hemorrhagic or thromboembolic events during peri-procedural period will be calculated globally and in each group (VKA or DOAC) as a percentage with 95% CI.

Financements Company's grant

* BMS
* DAIICHI SANKYO

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving long-term oral anticoagulant (defined as duration of treatment of at least 1 month) and referred for an invasive procedure (oral surgery, implantology or periodontology) to an oral surgeon member of the SFCO taking part to the study.

Each investigator will include 10 patients treated with long-term direct oral anticoagulants, and 10 consecutive patients treated with long-term Vitamin K Antagonists. For the oral anticoagulants group, inclusion will be continued until the inclusion of 333 patients for each molecule (apixaban, rivaroxaban, edoxaban).

Exclusion Criteria:

* Patients receiving both Vitamin K Antagonists and antiplatelet agents Patients receiving both direct oral anticoagulant and antiplatelet agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving oral anticoagulant undergoing an oral surgery, implantology or periodontology
Sampling Method: Non-Probability Sample
Enrollment: 532 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2017-07-04 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
The occurrence rate of bleeding or thromboembolic events during the peri-procedural period | Each patient will be followed for 30 days
  the occurrence rate of bleeding or thromboembolic events during the peri-procedural period defined as the period between 5 days before surgery plus 30 days after the invasive procedure (if no anticoagulant interruption) or 30 days after the resumption of oral anticoagulant (in case of an anticoagulant interruption).

SECONDARY OUTCOMES:
risk factors for bleeding in the peri-procedural period | Each patient will be followed for 30 days.
  To identify risk factors for bleeding in the peri-procedural period
risk factors for thromboembolic events in the peri-procedural period | Each patient will be followed for 30 days.
  To identify risk factors for thromboembolic events in the peri-procedural period
peri-procedural management of each treatment (VKA, and each DOAC) | Each patient will be followed for 30 days.
  To describe the peri-procedural management of each treatment (VKA, and each DOAC)
prescribers involved in the possible change of anticoagulant prescription prior the oral surgery | Each patient will be followed for 30 days.
  To identify prescribers involved in the possible change of anticoagulant prescription prior the oral surgery
risk of bleeding on DOAC and on VKA | Each patient will be followed for 30 days.
  To compare the risk of bleeding on DOAC and on VKA
risk of thromboembolic complications on DOAC and on VKA | Each patient will be followed for 30 days.
  To compare the risk of thromboembolic complications on DOAC and on VKA
net clinical benefit of DOAC compared to VKA treatment | Each patient will be followed for 30 days.
  To evaluate the net clinical benefit of DOAC compared to VKA treatment

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Mahé, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Louis Mourier, Colombes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Radoi L, Hajage D, Giboin C, Maman L, Monnet-Corti V, Descroix V, Mahe I. Perioperative management of oral anticoagulated patients undergoing an oral, implant, or periodontal procedure: a survey of practices of members of two dental scientific societies, the PRADICO study. Clin Oral Investig. 2019 Dec;23(12):4311-4323. doi: 10.1007/s00784-019-02877-1. Epub 2019 Mar 19. PMID 30887189